CLINICAL TRIAL: NCT00273741
Title: Randomized Study Evaluating the Antiasthenic Effect of Methylphenidate (Ritalin) in Palliative Care in Cancer Patients
Brief Title: Ritalin: Antiasthenic Effect of Methylphenidate (Ritalin) in Palliative Care in Cancer Patients
Acronym: Ritaline
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: difficulty of recrutement
Sponsor: University Hospital, Grenoble (Other)
Collaborators: Fondation de France (Other); Ligue contre le cancer, France (Other)
Responsible Party: Mr Marie, Direction de la recherche clinique et de l'innovation
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DCIC 03 29
Record Dates: First submitted 2006-01-06; First posted 2006-01-09 (Estimated); Last update posted 2009-12-07 (Estimated); Status verified 2009-12

CONDITIONS: Asthenia; Neoplasms
Keywords: palliative care; methylphenidate
MeSH Terms: conditions — Asthenia; Neoplasms | interventions — Methylphenidate; Exercise

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): methylphenidate at 20mg per day during 7 days, at 20mg or 40mg per day during 7 days and 20, 40 or 60mg per day during 14 days
  Interventions: Drug: methylphenidate
- 2 (Placebo Comparator): placebo capsules
  Interventions: Drug: placebo comparator

INTERVENTIONS:
Drug: methylphenidate — methylphenidate per os 20mg per day 7 days, 20mg or 40mg per day 7 days and 20, 40 or 60mg per day 14 days
  Other Names: active
  Arms: 1
Drug: placebo comparator — placebo capsules
  Other Names: placebo
  Arms: 2

SUMMARY:
The aim/objective of this study is to evaluate the antiasthenic effect of methylphenidate with a visual analogical scale (VAS) after 7 days of treatment, in cancer patients, in palliative care, i.e. with a progressive or terminal disease.

DETAILED DESCRIPTION:
Cancer patients in an advanced phase or who are terminally ill generally present with depression, pain, drowsiness, alterations of cognition, anorexia and other symptoms due to the progressive disease. The objective of the medical team of support and palliative care is to control these effects to maintain a quality of life. Particularly, the cancer patient in an advanced phase of the disease presents with important asthenia. In some patients, this asthenia is characterized by drowsiness or apathy. It always leads to ill-being and a sensation of bad adaptation. When an etiologic treatment is possible (correction of the anaemia, of the metabolic disorders, of the undernutrition, of the anorexia, of the insomnia, of the stubborn pain, of the psychological suffering), the asthenia can be fought. But, when it appears in patients not really in the end of life (life expectancy more than 1 month) and when no etiologic treatments are possible, other solutions must be considered, and all the more when the complaint is important with repeated requests for relief.

Methylphenidate is an amphetamine first indicated for deficient attention disorders with hyperactivity in children more than 6 years old. Several studies have been realized to evaluate its effect in cancer patients in palliative care. Some studies showed, in particular, its effectiveness on asthenia because of a stimulant and an antidepressant action. The methylphenidate could have an anti-analgesic effect or co-analgesic effect. All these studies are observational and not randomized. So they have a small level of proof and they have not been realized in a population of asthenic patients in palliative care. So a randomized controlled clinical trial in this specific population needs to be experimented.

ELIGIBILITY:
Inclusion Criteria:

* Advanced phase of neoplasm without any treatment available.
* Life expectancy of more than 1 month
* Karnofsky index more than 50%
* Chemotherapy IV or immunotherapy SC stopped more than 3 weeks before the end of the study
* Asthenia more than 5/10 on the visual analogical scale
* Informed consent form signed
* Affiliation to social security

Exclusion Criteria:

* Patients who can receive chemotherapy IV or immunotherapy SC in the month following the study
* Patients in whom disease can respond to chemotherapy
* Corticotherapy started less than 7 days before the study or potentially within the first week of the study
* Asthenia which can be easily corrected
* Contraindications to the amphetamines
* HADS score of anxiety and/or depression more than or egal to 17/21
* Potential surgery with general anesthesia in the first 7 days of the study
* Inability to quantify the sensation of asthenia on the visual analogical scale
* Pregnancy or feeding
* Guardianship

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2007-01; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Reduction of 3 units between the two study groups of the subjective impression of asthenia measured at the first day before the beginning of the treatment with a visual analogical scale at day 7 (+/- 1 day) | 7 days AVS

SECONDARY OUTCOMES:
Adverse events | each day
Visual analogical scale of pain | inclusion, day 1, 2, 3, 7, 14 and 28
European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ)-C30 | day 1, 7 and 28
Multidimensional Fatigue Inventory-20 (MFI-20) | day 1, 7, 14 and 28
Hospital Anxiety and Depression Scale (HADS) | inclusion, 7 and 28

CONTACTS AND LOCATIONS:
Overall Officials: Guillemette Laval, M.D., Ph.D., Principal Investigator — University Hospital, Grenoble
Locations (13):
- France (13):
  - Hôpital D'Annemasse, Annemasse
  - Centre Régional d'Accompagnement et de Soins Palliatifs,, Bordeaux
  - Equipe mobile de recherche et de soutien en soins pallitaifs, Grenoble
  - Unité de Soins palliatif, Centre Oscar Lambret, Lille
  - Unité de Soins Palliatifs, Hôpital Lyon sud, Lyon
  - Soins Palliatifs et Soins de support, Centre Léon Bérard, 28 rue Laënnec,, Lyon
  - Unité mobile de soutien et de soins palliatifs, Hôpital Saint-Eloi, Montpellier
  - EMSP, Institut Curie, Paris
  - EMSP, hôpital Saint aAntoine, Paris
  - Praz-Coutant, Passy
  - Unité de Soins Palliatifs, Saint-Etienne
  - EMSP, Hôpitaux du Léman, Thonon-les-Bains
  - Institut Gustave Roussy, Villejuif

REFERENCES:
- [Background] Bruera E, Miller MJ, Macmillan K, Kuehn N. Neuropsychological effects of methylphenidate in patients receiving a continuous infusion of narcotics for cancer pain. Pain. 1992 Feb;48(2):163-166. doi: 10.1016/0304-3959(92)90053-E. PMID 1589233
- [Background] Wilwerding MB, Loprinzi CL, Mailliard JA, O'Fallon JR, Miser AW, van Haelst C, Barton DL, Foley JF, Athmann LM. A randomized, crossover evaluation of methylphenidate in cancer patients receiving strong narcotics. Support Care Cancer. 1995 Mar;3(2):135-8. doi: 10.1007/BF00365854. PMID 7539701
- [Background] Rozans M, Dreisbach A, Lertora JJ, Kahn MJ. Palliative uses of methylphenidate in patients with cancer: a review. J Clin Oncol. 2002 Jan 1;20(1):335-9. doi: 10.1200/JCO.2002.20.1.335. PMID 11773187
- [Background] Bruera E, Chadwick S, Brenneis C, Hanson J, MacDonald RN. Methylphenidate associated with narcotics for the treatment of cancer pain. Cancer Treat Rep. 1987 Jan;71(1):67-70. PMID 3791269
- [Background] Bruera E, Driver L, Barnes EA, Willey J, Shen L, Palmer JL, Escalante C. Patient-controlled methylphenidate for the management of fatigue in patients with advanced cancer: a preliminary report. J Clin Oncol. 2003 Dec 1;21(23):4439-43. doi: 10.1200/JCO.2003.06.156. PMID 14645434